CLINICAL TRIAL: NCT05038566
Title: Dexterous Partial Hand Prosthesis Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Collaborators: Össur Iceland ehf (Industry)
Responsible Party: Principal Investigator, Todd Farrell, Director of Research, Liberating Technologies, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20212193
Record Dates: First submitted 2021-06-01; First posted 2021-09-09 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Amputation; Amputation; Traumatic, Hand; Limb; Absence, Congenital, Upper; Prosthesis User; Upper Limb Amputation at the Hand
Keywords: amputee; upper limb amputee; partial hand prosthesis user; prosthesis; i-Digits; upper limb loss; prosthetist; gripper; dexterous fingertip; index finger prosthesis

STUDY DESIGN:
Intervention Model Description: Functional tests will be used to evaluate the feasibility of the device design as compared with the subject's baseline device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Comparator Baseline (No Intervention): The subject's usual partial hand prosthesis
- Pointdexter (Experimental): The subject wears a modified version of their usual partial hand prosthesis. The modification replaces the usual index finger of the partial hand prosthesis with the investigational Pointdexter device.
  Interventions: Device: Pointdexter

INTERVENTIONS:
Device: Pointdexter — i-Digits partial hand prosthesis modified with the investigational pointdexter finger in place of the usual index finger.
  Other Names: Dexterous Partial Hand Prosthesis; Gripper
  Arms: Pointdexter

SUMMARY:
Liberating Technologies, Inc. (LTI) has developed a dexterous prosthetic fingertip that will be fit onto an i-Digits™ partial hand prosthesis and allow for an additional fine grasp. The device will interface with research participants' existing prostheses and use the same control strategy that is used for their everyday use. Each participant's prosthesis will be restored to their original configuration by the end of their testing period.

DETAILED DESCRIPTION:
Liberating Technologies, Inc. (LTI) has developed a dexterous prosthetic fingertip that will be fit onto an i-Digits™ partial hand prosthesis and allow for an additional fine grasp. The device will interface with research participant's existing prostheses and use the same control strategy that is used for their everyday use. Each participant's prosthesis will be restored to their original configuration by the end of their testing period.

The study will focus on design feasibility testing and will compare performance of hand functional outcome tests on an i-Digits™ prosthetic partial hand with and without the investigational Pointdexter modification. Our primary hypothesis is that subjects using the investigational device will show better performance on objective functional outcomes measures than those using a standard i-Digits™ partial hand prosthesis, particularly in the manipulation of small objects.

The investigators will explore multiple outcomes measures as options, but our primary endpoint will be performance on the Small Common Objects subtask of the Jebsen-Taylor Hand Function Test, which assesses a broad range of unimanual hand functions required for ADLs. The primary quantitative measure of the Jebsen-Taylor task will be completion time of each subtask. Qualitative evaluation will be conducted by an occupational therapist via observation, and by the user through a self-assessment questionnaire, such as the Patient Specific Functional Scale (PSFS). The investigators will be performing repeated measures on each individual subject to reduce the variance as well as having each subject act as their own control. New and existing i-Digits™ partial hand prosthesis users will be recruited for the study and consented with an approved protocol. Research participants will schedule a time to conduct the testing and be informed of study details.

The investigational device being tested is a novel prosthetic finger with a built-in split gripper. The device is an index finger which can drop in place of existing digits on an i-Digits™ partial hand prosthesis. The investigational device is controlled with the same signals as the conventional digits.

This study will pilot test the dexterous fingertip prosthesis with a small number of subjects (up to 12). Research participants will be consented and will test the device at home and/or in-lab. Subjects will be introduced to the partial hand prosthesis configuration and be instructed on how to operate it to complete their testing session.

The in-lab testing will be conducted in a single site visit at Össur Academy in Dublin, Ohio or LTI in Holliston, MA. Subjects may be asked to come back for an additional site visit if data collection is incomplete. For this study, the index finger of each participant's existing everyday prosthesis will be temporarily disconnected and replaced with the investigational device. The prosthesis will be restored to its original configuration when the test session has been completed. At the start of the study session, subjects will prepare for testing in their first configuration (investigational or comparator). If investigational, subjects will doff their prosthesis and investigators will replace the usual i-Digits™ index finger with the investigational device. If comparator, subjects will don their usual unmodified prosthesis. Subjects will be trained on how to operate the investigational device and be allowed a minimum of 30 minutes to practice using it until they are comfortable with proceeding. The subjects will be guided to conduct functional outcome tests that involve picking up and manipulating everyday objects (beans, coins, pegs, spoon, cloth, etc.), such as the tasks outlined in the Jebsen-Taylor and Peg Board functional tests. Each sub-task in the functional test will be scored by occupational therapist standards. After a round of functional testing is done, subjects will fill out the PSFS survey and subjective questionnaire. Subjects will then doff the prosthesis and don the next device configuration. The PSFS survey as well as user and clinician feedback are both exploratory outcome measures as the design is still in very early prototype stages. The intent of this feedback is to help iterate the design to assist in further development of the final product. Subjects will repeat the functional tests and surveys with each device configuration. After the final condition, the subject will have completed the study and their prosthesis will be restored to its usual configuration. The study session should span 3-5 hours.

A subset of subjects will take home the investigational device for up to 4 weeks to provide feedback of the device when used in everyday tasks. Investigators will restore the user's prosthesis at the end of the testing period and surveys will be conducted to capture feedback. Two site visits may be required: one to initialize the study and configure the prosthesis, and two to restore the prosthesis at the study end. This feedback is also an exploratory outcome measure due to the design being in very early prototype stages.

Both new and existing i-Digits™ partial hand prosthesis users will be invited to participate in the study. Research participants will schedule a time to conduct the testing and be informed of study details. Participants will be given as much time as needed to review and question the informed consent form before signing.

Two different technologies will be assessed:

* Investigational Device: i-Digits™ partial hand prosthesis with dexterous fingertip modification
* Comparator Baseline: unmodified i-Digits™ partial hand prosthesis

Persons with partial hand limb absence who are new or current i-Digits™ prosthesis users will be recruited for this study through the LTI and Össur clinician network. Prosthetists may be contacted with the need for research subjects and, if interested, will be given flyers to hand out to their patients. If subjects are interested in participating, they can call the number on the flyer to speak with investigators. In addition, previous research participants who have given permission to be contacted for future studies may be contacted directly to assess interest in participating in this study. Enrollment will be open to people of all ages, genders, races, and ethnicities. Participants must be new or current users of i-Digits™ partial hand prostheses. The user must have an absent index finger at minimum. Patients who have 4-5 digit and/or thumb involvement will be preferred.

Based on subject population and availability, a convenience sample of up to 12 subjects will be recruited for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Must have an upper limb partial hand absence.
* Must be new or current i-Digits prosthesis users.
* Must have an absent index finger at minimum.
* Must be able to understand spoken and written English in order to be properly consented and provide feedback to the study personnel.
* Must be willing and able to complete outlined tasks and provide feedback on the intervention.

Exclusion Criteria:

* The risks to pregnant women and fetuses are unknown and therefore pregnant women should not participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Farrell, PhD, Principal Investigator — Liberating Technologies, Inc.
Locations (2):
- United States (2):
  - Liberating Technologies, Inc., Holliston, Massachusetts
  - Össur Academy - Touch Solutions, Dublin, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Comparator Baseline, Then Pointdexter: The subject wears their usual partial hand prosthesis while performing functional outcome measures. The subject then wears a modified version of their usual partial hand prosthesis. The modification replaces the usual index finger of the partial hand prosthesis with the investigational Pointdexter device. Subjects will test out this hand configuration in the lab while performing functional outcome measures. This testing occurs at a single site visit (1 day) and lasts approximately 4 hours.
  Pointdexter: i-Digits partial hand prosthesis modified with the investigational pointdexter finger in place of the usual index finger.
- Pointdexter, Then Comparator Baseline: The subject wears a modified version of their usual partial hand prosthesis. The modification replaces the usual index finger of the partial hand prosthesis with the investigational Pointdexter device. Subjects will test out this hand configuration in the lab while performing functional outcome measures. The subject then wears their usual partial hand prosthesis while performing functional outcome measures. This testing occurs at a single site visit (1 day) and lasts approximately 4 hours.
  Pointdexter: i-Digits partial hand prosthesis modified with the investigational pointdexter finger in place of the usual index finger.
Period: Overall Study
Arm/Group | Comparator Baseline, Then Pointdexter | Pointdexter, Then Comparator Baseline
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Technical Difficulties with the Device | 0 | 1

BASELINE CHARACTERISTICS:
Population: Persons with partial hand amputation or partial hand difference with at least 4-5 digit involvement including the index finger.
Groups:
- Comparator Baseline, Then Pointdexter (~4 Hours of In-lab Testing): The subject wears their usual partial hand prosthesis while performing functional outcome measures. The subject then wears a modified version of their usual partial hand prosthesis. The modification replaces the usual index finger of the partial hand prosthesis with the investigational Pointdexter device. Subjects will either test out this hand configuration in the lab while performing functional outcome measures.
  The subject may then choose to take home the Pointdexter device for up to 4 weeks for feasibility testing of the early stage prototype device.
  Pointdexter: i-Digits partial hand prosthesis modified with the investigational pointdexter finger in place of the usual index finger.
- Pointdexter, Then Comparator Baseline (~4 Hours of In-lab Testing): The subject wears a modified version of their usual partial hand prosthesis. The modification replaces the usual index finger of the partial hand prosthesis with the investigational Pointdexter device. Subjects will test out this hand configuration in the lab while performing functional outcome measures. The subject then wears their usual partial hand prosthesis while performing functional outcome measures.
  The subject may then choose to take home the Pointdexter device for up to 4 weeks for feasibility testing of the early stage prototype device.
  Pointdexter: i-Digits partial hand prosthesis modified with the investigational pointdexter finger in place of the usual index finger.
- Total: Total of all reporting groups
Arm/Group | Comparator Baseline, Then Pointdexter (~4 Hours of In-lab Testing) | Pointdexter, Then Comparator Baseline (~4 Hours of In-lab Testing) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Jebsen-Taylor Small Common Objects Functional Test
Description: During the in-lab portion of the study, subjects will be asked to complete the 'small common objects' subtask of the Jebsen-Taylor Hand Function Test, which assesses a broad range of unimanual hand functions required for ADLs. The primary quantitative measure of the Jebsen-Taylor task will be completion time of each subtask. The maximum time allotted for each task was 120 seconds, at which point the subject was told to stop the task and the time was reported as the maximum 120 seconds. This test will be used to evaluate the feasibility of the device design as compared with a baseline condition.
  This was the only primary outcome measure collected for this study. There were no secondary outcome measures, only exploratory measures as this is a very early prototype design that is still in the design iteration stages.
Time Frame: 4 hours at a single site visit
Population: One participant was excluded from analysis due to an incomplete session because of technical difficulties with the device
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Comparator Baseline: The subject wears their usual partial hand prosthesis while performing functional outcome measures. Subjects will test out this hand configuration in the lab while performing functional outcome measures. This testing occurs at a single site visit (1 day) and lasts approximately 4 hours.
- Pointdexter: The subject wears a modified version of their usual partial hand prosthesis. The modification replaces the usual index finger of the partial hand prosthesis with the investigational Pointdexter device. Subjects will test out this hand configuration in the lab while performing functional outcome measures. This testing occurs at a single site visit (1 day) and lasts approximately 4 hours.
  Pointdexter: i-Digits partial hand prosthesis modified with the investigational pointdexter finger in place of the usual index finger.
Arm/Group | Comparator Baseline | Pointdexter
Number analyzed (Participants) | 2 | 1
Seconds
  Turning a Card Over | 34.8 (20.5) | 26.1 (4.5)
  Small Common Objects | 97.2 (32.2) | 62.1 (2.2)
  Stacking Checkers | 37.5 (43.1) | 28 (21.8)
  Manipulating Cloth | 5.4 (1.5) | 5.8 (1.7)
  Holding a Screw | 24.1 (1.8) | 65.7 (34.7)
  9-Hole Out | 11.4 (8.1) | 23.3 (19)
  9-Hole In | 120 (0) | 63.8 (57.3)
  Removing Pen Cap | 5.8 (2.3) | 7.1 (4.2)
  Tying Shoe Laces | 50.5 (49) | 34.6 (1.1)
  Zipping a Zipper | 32.6 (10.2) | 120 (0)
  Threading a Needle | 120 (0) | 32.4 (8.1)
  Simulated Feeding | 30.1 (22) | 66.3 (76)
  Large Light Objects | 11.7 (4.2) | 14.3 (3.7)
  Large Heavy Objects | 17.8 (4.6) | 16.7 (5)

ADVERSE EVENTS:
Time Frame: For the in-lab portion of the study, adverse events were monitored/assessed throughout the entire in-lab session, which was conducted over the course of 1 day. For the take-home early stage feasibility portion of the study, adverse events were monitored/assessed throughout the amount of time that subjects had the investigative device at home, which was up to 4 weeks.
Arm/Group | Comparator Baseline | Pointdexter
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT05038566/Prot_000.pdf